CLINICAL TRIAL: NCT01747512
Title: A Phase II/III Study of Cyclotron-produced Tc-99m Pertechnetate (C-PERT) Efficacy and Safety in Patients With Conformed and Suspected Thyroid Cancer or Head and Neck Cancer
Brief Title: An Imaging Study in Patients With Thyroid Cancer or Head and Neck Cancer With Pertechnetate Made in a Cyclotron (C-PERT)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was not initiated
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DX-CPERT-002
Record Dates: First submitted 2012-12-10; First posted 2012-12-11 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Thyroid Neoplasms; Head and Neck Neoplasms
Keywords: 99mTc Pertechnetate; thyroidectomy; thyroid neoplasms
MeSH Terms: conditions — Thyroid Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- C-PERT (Active Comparator): 45 patients with cancer
  Interventions: Drug: C-PERT
- G-PERT (Active Comparator): 65 patients with cancer
  Interventions: Drug: G-PERT

INTERVENTIONS:
Drug: C-PERT — Patients with thyroid and Head and Neck cancer
  Arms: C-PERT
Drug: G-PERT — Patients with thyroid and Head and Neck cancer
  Arms: G-PERT

SUMMARY:
Doctors at the Cross Cancer Institute have developed a new method of producing 99mTc Pertechnetate in a cyclotron unit. A study done at the Cross Cancer Institute in 2011 with ten patients using this imaging agent showed that it was safe and produced images with the same pattern as generator produced Pertechnetate. This study is now being done in larger numbers of patients to again show that the imaging pattern of both agents is the same, and to again demonstrate its safety.

DETAILED DESCRIPTION:
To demonstrate the efficacy of cyclotron-produced Tc-99m pertechnetate (C-PERT; manufactured by the Edmonton PET Centre/ERC) in comparison to generator-produced Tc-99m pertechnetate (G-PERT; from approved commercial source; using qualitative and quantitative clinical imaging biodistribution data.

ELIGIBILITY:
Inclusion Criteria:

* thyroid cancer, or
* Head and Neck cancer for salivary gland transfer
* age 18-79
* biochemical parameters < 5x ULN
* WBC > 3.0/uL
* ANC > 1.5/uL
* platelets > 75,000/uL
* hemoglobin > 10 g/dL
* Karnofsky 50-100

Exclusion Criteria:

* nursing or pregnant females
* < 18 or > 79 Years
* uncontrolled asthma
* acute iritis
* narrow angle glaucoma
* previous radiation to head/neck

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the efficacy of C-PERT (manufactured by the Edmonton PET Centre/ERC) in comparison to G-PERT (fromm approved commercial sources) using qualitative and quantitative clinical imaging biodistribtion data. | 5 months

SECONDARY OUTCOMES:
To evaluate the safety of C-PERT from adverse event data | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Alexander McEwan, MB, FRCPC, Principal Investigator — Professor, Department of Oncology